CLINICAL TRIAL: NCT05193318
Title: Ketamine-assisted Psychotherapy for the Treatment of Persistent Depression in Abstinent Opioid Users
Brief Title: KAP for Depression in Abstinent Opioid Users
Acronym: KReDO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Investigator leaving institution
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Eric Dobson, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115696
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use Disorder, Severe, in Sustained Remission; Opioid Use Disorder, Severe, in Early Remission; Major Depressive Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine-assisted psychotherapy (Experimental): Subjects will receive 8 weekly intramuscular injections of ketamine hydrochloride starting at 0.5 mg/kg and increasing to a maximum dose of 1.5 mg/kg or a total dose of 60 mg, whichever is lower. Ketamine administration will be accompanied by psychotherapy before, after and during the session.
  Interventions: Drug: Ketamine-assisted psychotherapy

INTERVENTIONS:
Drug: Ketamine-assisted psychotherapy — Subjects will receive 8 weekly intramuscular injections of ketamine hydrochloride starting at 0.5 mg/kg and increasing to a maximum dose of 1.5 mg/kg or a total dose of 60 mg, whichever is lower. Ketamine administration will be accompanied by psychotherapy before, after and during the session.

SUMMARY:
The purpose of the study is to examine whether an investigational medication called ketamine along with psychotherapy is an effective treatment for depression in participants with a history of opioid addiction who have not abused opioids in at least 3 months. Participants will receive ketamine through intramuscular injection along with psychotherapy weekly for 8 weeks. Participation for eligible subjects who decide to enroll (including post-medication follow-up visits) will last about 16 weeks or 4 months.

ELIGIBILITY:
Inclusion Criteria

A subject may be eligible for enrollment if all the following inclusion criteria apply within the thirty days prior to first experimental session:

1. Between the ages of 18 to 64 years old.
2. Able to provide informed consent.
3. Meet DSM-5 criteria for Major Depressive Disorder, without psychotic features based on clinical interview.
4. Score at least 20 on the Montgomery-Asberg Depression Rating Scale (MADRS, moderate or severe depression).
5. Must meet criteria for opioid use disorder in early or sustained remission criteria by DSM-5 based on clinical interview.
6. Subjects taking other psychotropic medications (e.g. anti-depressants, anxiolytics, methadone, buprenorphine, naltrexone) must be maintained on a stable dose for at least four weeks before study initiation.

Exclusion Criteria

Subjects will be excluded from the study if any of the following criteria apply:

1. They are considered an immediate suicide risk by clinician assessment, self-reports a suicide attempt within the past year, or felt to be likely to require hospitalization during the study.
2. Subjects who meet DSM-5 criteria for current bipolar disorder based on clinical interview.
3. Subjects who meet DSM-5 criteria for current or history of psychotic spectrum disorders based on clinical interview.
4. Subjects meeting DSM-5 criteria for current substance use disorder (i.e., not in early or sustained remission) other than tobacco use disorder.
5. Subjects who report use of ketamine >20 times in the past or who meet DSM-5 criteria for Other Hallucinogen Use Disorder due to ketamine use including subjects who are currently in early or sustained remission.
6. Women who are pregnant or nursing, and women who do not consent to use methods of highly effective birth control during the interventional phase of the study.
7. Subjects with hypertension as defined by a baseline visit systolic blood pressure (SBP) >140 mmHg or a diastolic blood pressure (DBP) >90 mmHg.
8. A history of allergic or other adverse reaction to ketamine (or its excipients).
9. Clinically significant physical exam findings or self-reported medical conditions for which a transient increase in blood pressure could be significantly detrimental (e.g. glaucoma, aneurysmal disease, cardiovascular disease, or end-stage renal disease).
10. QTc will be measured in all subjects and those with QTc 450ms or longer will be excluded.
11. Subjects who live greater than 20 miles from the study site and cannot arrange their own transportation will be excluded from the study.
12. Subjects with kidney or liver impairment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Dobson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Centerspace, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intended total recruitment was 10 participants, however study was concluded after a total of 5 participants were recruited.
Period: Acute Intervention (Weeks 1-9 of Study)
Arm/Group | Ketamine-assisted Psychotherapy
Started | 5
Completed | 4
Not Completed | 1
Not completed — Physician Decision | 1
Period: Follow-up Phase (Through Week 16)
Arm/Group | Ketamine-assisted Psychotherapy
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Sexual orientation [Count of Participants; unit: Participants]
  Heterosexual | 3
  Homosexual | 1
  Bisexual | 1
MADRS baseline [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS). The MADRS is a clinician administered, 10-item questionnaire of depression severity. The total score ranges from 0-60, with scores of 0-6 considered normal (non-depressed), 7-19 indicative of mild depression, 20-34 indicative of moderate depression, and 35-60 indicative of severe depression. Lower scores are better (less depressed).
  units on a scale | 34.0 (6.0)
BDI Baseline [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory (BDI-II). A widely used 21-item self-report measure of depressive symptoms. The range of possible scores is 0 to 63. BDI-II scores are classified as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63). Lower scores are better (less depressed).
  units on a scale | 42.8 (7.7)
GAD-7 Baseline [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder Screener (GAD-7). The GAD-7 is a 7-item self report instrument that will assess generalized anxiety symptomatology. Total range is 0-21. GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe). Lower scores are better (less anxious).
  units on a scale | 18.4 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale
Description: Montgomery Asberg Depression Rating Scale (MADRS). The MADRS is a clinician administered, 10-item questionnaire of depression severity. The total score ranges from 0-60, with scores of 0-6 considered normal (non-depressed), 7-19 indicative of mild depression, 20-34 indicative of moderate depression, and 35-60 indicative of severe depression. Individuals scoring 20 or higher on the MADRS will be included in the study. The MADRS evaluates the following symptoms of depression: 1) clinical appearance of sadness, 2) self-reported sadness, 3) inner tension, 4) reduced sleep, 5) reduced appetite, 6) concentration difficulties, 7) lassitude, 8) inability to feel, 9) pessimistic thought process, and 10) thoughts of suicide. Lower scores are better (less depression).
Time Frame: Change from baseline measured at week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 16
Population: Includes participants with available data. One participant dropped out after week 2, another failed to follow-up after week 9.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Week 1 | -1.75 (3.5)
  Week 2 | -3.25 (3.0)
  Week 3: number analyzed (Participants) | 4
  Week 3 | -7.25 (7.27)
  Week 4: number analyzed (Participants) | 4
  Week 4 | -11.75 (7.37)
  Week 5: number analyzed (Participants) | 4
  Week 5 | -9 (6.98)
  Week 6: number analyzed (Participants) | 4
  Week 6 | -18.3 (6.18)
  Week 7: number analyzed (Participants) | 4
  Week 7 | -19 (4.83)
  Week 8: number analyzed (Participants) | 4
  Week 8 | -20 (6.32)
  Week 9: number analyzed (Participants) | 4
  Week 9 | -15.5 (7.55)
  Week 10: number analyzed (Participants) | 3
  Week 10 | -10.7 (12.7)
  Week 12: number analyzed (Participants) | 3
  Week 12 | -8.33 (18.15)
  Week 16: number analyzed (Participants) | 3
  Week 16 | -10.67 (15.82)

2. Secondary Outcome: Beck Depression Inventory
Description: Self-rated depression inventory; minimum score of 0 maximum score of 63 with lower scores being a better outcome (less depressed)
Time Frame: Change from baseline measured at week 1-9, 10, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Week 1 | -1.6 (1.7)
  Week 2 | -6.4 (5.0)
  Week 3: number analyzed (Participants) | 4
  Week 3 | -8.8 (11.3)
  Week 4: number analyzed (Participants) | 4
  Week 4 | -11.8 (9.8)
  Week 5: number analyzed (Participants) | 4
  Week 5 | -9 (12.2)
  Week 6: number analyzed (Participants) | 4
  Week 6 | -13 (9.1)
  Week 7: number analyzed (Participants) | 4
  Week 7 | -15.5 (8.5)
  Week 8: number analyzed (Participants) | 4
  Week 8 | -18 (9.6)
  Week 9: number analyzed (Participants) | 4
  Week 9 | -17.3 (10.3)
  Week 10: number analyzed (Participants) | 3
  Week 10 | -15.3 (9.5)
  Week 12: number analyzed (Participants) | 3
  Week 12 | -13.7 (16.3)
  Week 16: number analyzed (Participants) | 3
  Week 16 | -16.7 (9.9)

3. Secondary Outcome: Visual Analog Scale (VAS)
Description: Measure of subjective level of opioid craving; maximum score of 100 and minimum score of 0 with higher scores meaning worse outcome (more cravings)
Time Frame: Change relative to baseline measured at week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Week 1 | 5 (17.97)
  Week 2 | 5 (37.3)
  Week 3: number analyzed (Participants) | 4
  Week 3 | 9.25 (43.14)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 4.75 (47.77)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 10 (49.48)
  Week 6: number analyzed (Participants) | 4
  Week 6 | -1.25 (38.43)
  Week 7: number analyzed (Participants) | 4
  Week 7 | -1.75 (33.09)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 1.25 (36.55)
  Week 9: number analyzed (Participants) | 4
  Week 9 | -6 (38.17)
  Week 10: number analyzed (Participants) | 3
  Week 10 | -2 (55.03)
  Week 12: number analyzed (Participants) | 3
  Week 12 | -4.33 (54.63)
  Week 16: number analyzed (Participants) | 3
  Week 16 | -11 (42.58)

4. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: Self-report of anxiety symptom severity; minimum score of 0 and maximum score of 21 with higher scores meaning worse outcome (more anxious)
Time Frame: Change in score relative to baseline calculated at week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 16.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Week 1 | -2.2 (3.35)
  Week 2 | -4.2 (3.11)
  Week 3: number analyzed (Participants) | 4
  Week 3 | -6.75 (4.72)
  Week 4: number analyzed (Participants) | 4
  Week 4 | -6.5 (3.11)
  Week 5: number analyzed (Participants) | 4
  Week 5 | -6.25 (3.59)
  Week 6: number analyzed (Participants) | 4
  Week 6 | -8.75 (4.43)
  Week 7: number analyzed (Participants) | 4
  Week 7 | -7 (5.03)
  Week 8: number analyzed (Participants) | 4
  Week 8 | -9 (3.37)
  Week 9: number analyzed (Participants) | 4
  Week 9 | -8.75 (4.92)
  Week 10: number analyzed (Participants) | 3
  Week 10 | -6.33 (4.16)
  Week 12: number analyzed (Participants) | 3
  Week 12 | -8.33 (6.11)
  Week 16: number analyzed (Participants) | 3
  Week 16 | -9 (5)

5. Secondary Outcome: Mystical Experience Questionnaire (MEQ)
Description: Measure of perceptual experiences; multiple items rated on a 5 point scale with higher scores indicating more intense perceptual experience. Total scores are presented as an average (mean) of the 30 item scale, each of which are rated out of 5. Scale is ordered as follows (in reference to magnitude of various perceptual experiences during acute ketamine session): 0 - none; not at all; 1 - so slight cannot decide; 2 - slight; 3- moderate; 4 - strong (equivalent in degree to any other strong experience); 5- extreme (more than any other time in my life and stronger than 4).
Time Frame: Measured at week 1-8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Week 1 | 2.96 (1.20)
  Week 2 | 2.32 (1.37)
  Week 3: number analyzed (Participants) | 4
  Week 3 | 3.55 (0.81)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 3.54 (0.81)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 3.88 (0.87)
  Week 6: number analyzed (Participants) | 4
  Week 6 | 3.25 (0.84)
  Week 7: number analyzed (Participants) | 4
  Week 7 | 4.28 (0.55)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 3.9 (0.78)

6. Secondary Outcome: Brief Pain Inventory (BPI)
Description: Measure of pain. Sub-scale 3 specifically was reported for this outcome. Subjects were asked: "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last 24 hours"; maximum score of 10 and minimum of 0 with higher scores indicating worse outcome (more pain) and a score of 0 indicating best outcome (no pain).
Time Frame: Measured at baseline, week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
score on a scale
  Baseline | 1.4 (1.95)
  Week 1 | 1.6 (2.30)
  Week 2 | 1.2 (2.17)
  Week 3: number analyzed (Participants) | 4
  Week 3 | 0.33 (0.58)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 0 (0)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 0 (0)
  Week 6: number analyzed (Participants) | 4
  Week 6 | 0 (0)
  Week 7: number analyzed (Participants) | 4
  Week 7 | 0 (0)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 0 (0)
  Week 9: number analyzed (Participants) | 4
  Week 9 | 0 (0)
  Week 10: number analyzed (Participants) | 3
  Week 10 | 0 (0)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 0 (0)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 0 (0)

7. Secondary Outcome: PTSD Checklist (PCL-5; PTSD Checklist 5)
Description: Measure of PTSD symptoms; maximum score 80 and minimum score of 0 with higher scores indicating worse outcome (more PTSD symptoms)
Time Frame: Measured at week 1-9, 10, 12, and 16
Population: Includes participants with available data. Four patient endorses trauma and completed PCL at least once. One participant inconsistently endorsed trauma depending on assessment week, leading to variation in number of participants analyzed each week. One participant dropped out after week 2, another failed to follow-up after week 9.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 4
score on a scale
  Week 1: number analyzed (Participants) | 3
  Week 1 | 64 (7.55)
  Week 2 | 54 (17.08)
  Week 3: number analyzed (Participants) | 3
  Week 3 | 42.33 (19.09)
  Week 4: number analyzed (Participants) | 3
  Week 4 | 45.33 (18.04)
  Week 5: number analyzed (Participants) | 2
  Week 5 | 44 (21.21)
  Week 6: number analyzed (Participants) | 3
  Week 6 | 32.33 (18.93)
  Week 7: number analyzed (Participants) | 2
  Week 7 | 37 (31.11)
  Week 8: number analyzed (Participants) | 2
  Week 8 | 36 (19.80)
  Week 9: number analyzed (Participants) | 2
  Week 9 | 37 (25.46)
  Week 10: number analyzed (Participants) | 2
  Week 10 | 40.5 (28.99)
  Week 12: number analyzed (Participants) | 2
  Week 12 | 39 (33.94)
  Week 16: number analyzed (Participants) | 2
  Week 16 | 38.5 (27.58)

8. Secondary Outcome: Timeline Follow-back (TLFB)
Description: Measure of Substance Use; maximum number of substance use days per week is 7 and minimum is 0 with higher number indicating worse outcomes (more substance use)
Time Frame: Measured at week 1-9, 10, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Ketamine-assisted Psychotherapy
Number analyzed (Participants) | 5
days per week
  Week 1 | 0.6 (1.34)
  Week 2 | 0 (0)
  Week 3: number analyzed (Participants) | 4
  Week 3 | 0 (0)
  Week 4: number analyzed (Participants) | 4
  Week 4 | 0 (0)
  Week 5: number analyzed (Participants) | 4
  Week 5 | 1 (2)
  Week 6: number analyzed (Participants) | 4
  Week 6 | 0.35 (0.7)
  Week 7: number analyzed (Participants) | 4
  Week 7 | 0 (0)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 0 (0)
  Week 9: number analyzed (Participants) | 4
  Week 9 | 0 (0)
  Week 10: number analyzed (Participants) | 3
  Week 10 | 0 (0)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 0 (0)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 0 (0)

ADVERSE EVENTS:
Time Frame: 16 weeks after initiation of acute intervention
Arm/Group | Ketamine-assisted Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine-assisted Psychotherapy (N=5)
Nausea (Gastrointestinal disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05193318/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT05193318/ICF_001.pdf